CLINICAL TRIAL: NCT03706729
Title: Fear of Re-injury and Ankle Function in Elite Athletes With Chronic Ankle Instability Using the Spraino® Shoe Patch: A Cohort Study
Brief Title: Elite Athletes With Chronic Ankle Instability Using Spraino®: A Cohort Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Covid-19 pandemic
Sponsor: University of Southern Denmark (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other); Aalborg University (Other); Metropolitan University College (Other); Spraino (Industry)
Responsible Party: Principal Investigator, Behnam Liaghat, Principal Investigator, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SprainoCohortStudy
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Chronic Ankle Instability
Keywords: Ankle injury; Joint instability; Prevention and control; Elite athletes; Indoor Sports; Ligamentous sprain; Fear of re-injury
MeSH Terms: conditions — Ankle Injuries; Joint Instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spraino intervention group (Experimental): Participants will use Spraino® as a measure to prevent future lateral ankle sprains during all training sessions and games.
  Interventions: Device: Spraino

INTERVENTIONS:
Device: Spraino — Spraino® is an adhesive polytetrafluoroethylene (PTFE or "Teflon") patch developed with the purpose of minimizing lateral shoe-surface friction whenever initial contact is carried out in an inverted position of the ankle joint. Each Spraino® PTFE patch has a minimum durability of 20 hours use and will be provided by the study sponsor, Spraino® ApS. The participants will receive four pairs of Spraino® upon their enrollment to the study.

SUMMARY:
Fear of re-injury and deficiencies in ankle joint function are common conditions amongst high performance (elite) athletes with chronic ankle instability (CAI), who participate in indoor sports. This fear of re-injury associates with the high recurrence rate of lateral ankle sprains, which is a primary characteristic feature of CAI. The Spraino® shoe patch is a new Danish invention, which is designed to reduce the risk of sustaining lateral ankle sprains in this population. This cohort study will investigate self-reported fear of re-injury and objectively measured ankle joint function in elite indoor sports athletes with CAI, both before and after a 10-week period during which they will use Spraino® during all training sessions and games.

DETAILED DESCRIPTION:
Acute lateral ankle sprains are frequently incurred by athletes, who participate in indoor sports such as volleyball, handball, and badminton; accounting for up to 30% of all injuries sustained in these sports. Despite established injury prevention strategies, the prevalence of recurrent lateral ankle sprain injuries and the concomitant development of CAI is high for athletes participating in indoor sports. CAI is characterized by athlete self-reported feelings of ankle joint instability, episodes of ankle joint "giving-way", and recurrent lateral ankle sprains. Additionally, athletes with CAI, who participate in indoor sports, may develop a heightened fear of re-injury, which may deter them from performing optimally in their sport. This study is designed as a prospective cohort study. The objective is to investigate fear of re-injury and ankle function in elite athletes with CAI (n = 25), both before and after a 10-week period during which they will use Spraino® during all training sessions and games. This study seeks to answer the following research questions: Does fear of re-injury improve in elite indoor sports athletes with established CAI when using Spraino® for 10 weeks? Does the use of Spraino® improve their ankle function?

The intervention time is scheduled for 10 weeks with the primary time point of interest being at the completion of week 10. The combined number of training sessions and games for each participant over the 10-week time-period is anticipated to exceed 32 exposures to ensure adequate exposure of participants to the use of Spraino®. All participants will receive a weekly text message using a Short Message Services-system (SMS-Track) throughout the 10-week time-period. This will be used to quantify training and game exposure and to register occurrences of new ankle injuries.

Embedded in this study is a qualitative method (semi-structured interview after week 10) to assess the participants´ experiences of using Spraino®. The content analysis will be a descriptive analysis of the data with some degree of interpretive analysis. The qualitative study will be reported in a secondary paper with a clear reference to this primary study registration.

The study purpose and methodology were evaluated by four identified stakeholders from the highest sports level including a physiotherapist, a head coach, a team doctor and an athlete. Their feedback ensured that the research is relevant to real-life circumstances and adds value to existing injury prevention strategies in elite indoor team sport.

The enrollment process will start in October 2018 and conclude when 25 participants have been enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥ 18 years old at commencement of study.
* Participant can read, speak and understand English.
* Participant is playing in one of the two highest leagues in the following indoor sports: handball, volleyball and badminton with at least 32 training sessions during the study period.
* Participant is diagnosed with CAI using the definition endorsed by the International Ankle Consortium.:

  * Participant has previously incurred at least one significant lateral ankle sprain that resulted in swelling, pain, and temporary loss of function at least 12 months prior to study enrollment.
  * Participant has a history of multiple episodes of the ankle ''giving-way'', and/or recurrent sprain and/or "feelings of instability" in the past six months
  * Participant has a Cumberland Ankle Instability Tool (CAIT) score <24
* Participant can fully participate in training sessions and is eligible for game selection before enrollment in the study.
* Participant can receive and reply to text messages on a cell phone using Short Message Services (SMS).

Exclusion Criteria:

* History of medial ankle sprain
* History of ankle surgery
* Participant who does not agree to sign the informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Fear of re-injury (Continuous) | 10 weeks
  Fear of re-injury will be measured using a Numeric Rating Scale (NRS) from 0 to 100 with 10-point increments (e.g. by asking the participants: "How fearful are you of re-injuring your ankle?"), with lower scores indicating more fear of re-injury.

SECONDARY OUTCOMES:
Y-balance test (Continuous) | 10 weeks
  The athletes must maintain single-leg balance on one leg while reaching as far as possible with the contralateral leg in three different directions, including anterior, posteromedial and posterolateral performed on each leg. The test measures a reaching distance (normalized to percentage of the leg length) on the M.A.T (Movement Assessment Technologies) system.
  After completion of the test, three self-reported questions will be administered regarding pain, how confident and how stable the participants feel in their ankle. Score ranges from 0 (no pain/ fully confident/ fully stable) to 10 (worst possible pain/not at all confident/ not at all stable) on an 11-point NRS.
The side-hop test (fastest time). (Continuous) | 10 weeks
  The athletes must hop on one leg laterally and back again over a 30-cm distance (counted as one repetition). The test measures the time (seconds) it takes to complete 10 repetitions.
  After completion of the test, three self-reported questions will be administered regarding pain, how confident and how stable the participants feel in their ankle. Score ranges from 0 (no pain/ fully confident/ fully stable) to 10 (worst possible pain/not at all confident/ not at all stable) on an 11-point NRS.
The Foot and Ankle Ability Measure (FAAM) sports scale | 10 weeks
  The Foot and Ankle Ability Measure (FAAM) sports scale is an 8-item questionnaire designed to assess the level of ankle function in sports. Each item is scored on a five-point Likert scale from 4 to 0. Total scores can vary from 0 to 32, with higher scores representing higher levels of physical function.
Tampa Scale of Kinesiophobia-11 (TSK-11) | 10 weeks
  The Tampa Scale of Kinesiophobia-11 (TSK-11) is an 11-item questionnaire designed to assess fear of movement and re-injury. All items are based on a 4-point Likert scale in which athlete options range from strongly disagree to strongly agree. The TSK-11 scores range from 11 to 44, with higher scores indicating more kinesiophobia.
Fear-Avoidance Beliefs Questionnaire (FABQ) | 10 weeks
  The FABQ is a 16-item questionnaire designed to assess fear-avoidance beliefs. Each item is scored on a 7-point Likert scale from completely disagree to completely agree. The FABQ scores range from 0 to 66, with higher scores representing increased fear-avoidance beliefs.
Time-loss due to an ankle sprain | 10 weeks
  Time-loss (in days) due to an ankle sprain per athlete (continuous)
The athlete experience with Spraino® (qualitative) | 10 weeks
  Semi-structured interview regarding the participants´experiences from using Spraino® as preventative measure

OTHER OUTCOMES:
Registration of adverse effects | 10 weeks
  Adverse effects from using Spraino® (Binary) The participants will be encouraged to report occurrences of adverse events related to their use of Spraino® to the primary investigator. These events will be registered and reported to the Ethical Committee within seven days.

CONTACTS AND LOCATIONS:
Overall Officials: Behnam Liaghat, MSc, Principal Investigator — Department of Sports Science & Clinical Biomechanics, University of Southern Denmark, Odense, Denmark; Kristian Thorborg, PhD, Study Director — Physical Medicine and Rehabilitation Research-Copenhagen (PMR-C), Clinical Research Centre, Amager-Hvidovre Hospital, Copenhagen University, Hvidovre, Denmark; Thomas Q Bandholm, PhD, Study Chair — Physical Medicine and Rehabilitation Research-Copenhagen (PMR-C), Clinical Research Centre, Amager-Hvidovre Hospital, Copenhagen University, Hvidovre, Denmark; Eamonn Delahunt, PhD, Study Chair — School of Public Health, Physiotherapy and Sports Science, University College Dublin, Dublin, Ireland
Locations (2):
- Denmark (2):
  - Physical Medicine and Rehabilitation Research-Copenhagen (PMR-C), Clinical Research Centre, Amager-Hvidovre Hospital, Copenhagen University, Hvidovre
  - Department of Sports Science and Clinical Biomechanics, University of Southern Denmark, Odense, Denmark, Odense

IPD SHARING:
Plan to Share IPD: Undecided